CLINICAL TRIAL: NCT04033055
Title: Interventional Study of Antalgic Efficacy of the CycloMesh™ Implant Soaked in Ropivacaine Hydrochloride 10 Mg/mL in the Treatment of Uncomplicated Inguinal Hernia. Randomized Comparative Study Versus CycloMesh™ Soaked in Physiological Saline Solution NaCl 9°/°°
Brief Title: Antalgic Efficacy of CycloMesh™ Soaked in Ropivacaine Hydrochloride in Uncomplicated Inguinal Hernia.
Acronym: HENRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2891
Record Dates: First submitted 2019-07-15; First posted 2019-07-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient will be blinded to the randomisation arm. As the procedure is conducted under general anaesthesia, the patient will not be informed whether the procedure which was performed on him/her did or did not result in the implantation of the CycloMesh™ device. Also, the surgeon such as the outcome assessor will be blinded to the randomisation arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CycloMesh™ soaked in ropivacaine hydrochloride 10mg/mL (Experimental): The surgical technique for the inguinal hernia repair is the surgeon's usual technique: open surgery (Lichtenstein technique).
  CycloMesh™ device (soaked in ropivacaine hydrochloride 10mg/mL) is positioned once the surgery for the inguinal hernia repair has been performed.
  Interventions: Procedure: Inguinal hernia repair with CycloMesh™ soaked in ropivacaine hydrochloride 10mg/mL
- CycloMesh™ soaked in saline solution 9°/°° (Active Comparator): The surgical technique for the inguinal hernia repair is the surgeon's usual technique: open surgery (Lichtenstein technique).
  CycloMesh™ device (soaked in saline solution) is positioned once the surgery for the inguinal hernia repair has been performed.
  Interventions: Procedure: Inguinal hernia repair with CycloMesh™ soaked in saline solution NaCl 9°/°°

INTERVENTIONS:
Procedure: Inguinal hernia repair with CycloMesh™ soaked in ropivacaine hydrochloride 10mg/mL — The surgical technique for the inguinal hernia repair is the surgeon's usual technique: open surgery (Lichtenstein technique).
  CycloMesh™ device (soaked in ropivacaine hydrochloride 10mg/mL) is positioned once the surgery for the inguinal hernia repair has been performed.
  Arms: CycloMesh™ soaked in ropivacaine hydrochloride 10mg/mL
Procedure: Inguinal hernia repair with CycloMesh™ soaked in saline solution NaCl 9°/°° — The surgical technique for the inguinal hernia repair is the surgeon's usual technique: open surgery (Lichtenstein technique).
  CycloMesh™ device (soaked in saline solution) is positioned once the surgery for the inguinal hernia repair has been performed.
  Arms: CycloMesh™ soaked in saline solution 9°/°°

SUMMARY:
CycloMesh is a polyester visceral implant functionalized by drug delivery systems directly on its surface, targeting a unique intervention, a slow anesthetic release and an in situ activity. Based on the fact that cyclodextrins are capable of forming inclusion complexes with amino-amide anaesthetic agents, ropivacaine and cyclodextrins were combined on a commercial visceral mesh.This enables CycloMesh to release ropivacaine for a sustained period in order to improve patient's comfort after inguinal hernia surgery.

The underlying hypothesis of this work is that clinical gain is achieved by adding a drug delivery system to visceral mesh for the local and prolonged delivery of ropivacaine. This should results in an improvement in quality of life, a reduction in pain and a faster returning to work following treatment of inguinal hernia by lichtenstein technique.

ELIGIBILITY:
Inclusion Criteria:

Disease-related criteria:

* Uncomplicated and non-recurrent unilateral symptomatic inguinal hernia with a surgical indication
* Bilateral inguinal hernia symptomatic on one side and requiring surgery on the symptomatic side
* Symptomatic, normal unilateral inguino-scrotal hernia (located above the middle of the inner thigh), uncomplicated and non-recurrent, with an indication for surgery by local inguinal approach without testicular redonation.
* Open surgery with Lichtenstein's technique;
* Programmed outpatient surgery;
* Surgery performed under general anesthesia.

Population-related criteria:

* Male subjects over 18 years old;
* Subjects who have given their free informed signed consent to participate in the study;
* Subjects who are affiliated to a social security system or have rights from a social security system.

Non inclusion Criteria:

Disease-related criteria:

* Strangulated inguinal or inguino-scrotal hernia;
* Bilateral inguinal hernia symptomatic on both sides and requiring surgery on both sides
* Chronic pain state (> 3 months) and/or long term analgesics intake susceptible to hide or interfere with pain assessment;
* Hepatic or renal failure and any other pathology that could notably extend half-life of anaesthetics and analgesics products
* Signs of infection at the surgical site;
* Severe cardiopulmonary, hepatic or renal diseases
* Active ongoing malignant disease;

Product or device-related criteria:

* Known allergy or hypersensitivity to any of the constituents of the CycloMesh (Polyethylene terephthalate + Cyclodextrin) and/or subjects allergic to ropivacaine;
* Allergy to any drugs of the anesthesia protocol;

Population-related criteria:

* Drug or alcohol abuse (addiction: i.e. chronic alcoholism or active drug addiction)
* Daily intake of level I analgesics (Paracetamol, Aspirin, Ibuprofen...etc.), for > 6 weeks.
* Use of corticosteroids within 24 hours prior to the surgery.
* Chronic use of antidepressants, anxiolytics, neuroleptics since 1 month or more,
* In case of occasional use, taking antidepressants, anxiolytics, neuroleptics in the 72 h prior to the intervention
* Unavailability during the study
* Participation in a clinical trial within 3 months prior to the initial visit.
* Psychiatric pathology or depressive disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity after treatment of inguinal hernia by lichtenstein technique under general anesthetic will be assessed 6h post-operative using Visual Analogic Scale (VAS). | 6 hours post-surgery
  The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate. It is a self-assessment scale and is sensitive, reproducible, reliable and validated for both acute and chronic pain situations.
  Pain assessment will be performed 6 hours after implant placement and during cough effort.

SECONDARY OUTCOMES:
Pain intensity back to home (Day 0) and Day 1 to 3 will be assessed using a Visual Analogic Scale (VAS) | Back to home (Day 0) at 8pm and 10 pm, Twice a day (8 am and 8 pm) at Day 1, Day 2 and Day 3
  Pain intensity will be reported by the patient on a log book using a Visual Analogic Scale . The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate
Pain intensity at Day 1 and Day 7 post-surgery will be assessed using a Visual Analogic Scale (VAS) | Day 1 and Day 7 post-surgery
  Pain intensity at Day 1 and Day 7 post-surgery will be assessed using a visual analogic scale and during a telephone interview performed by an investigator's collaborator.
  The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate.It is a self-assessment scale and is sensitive, reproducible, reliable and validated both in acute pain and chronic pain situations.
Pain intensity at 1 month post-surgery will be assessed using a Visual Analogic Scale (VAS) | 1 month post-surgery
  Pain intensity at 1 month post-surgery will be assessed, using a visual analogic scale, during a visit to the surgeon and in 3 different situations: at rest, walking and during cough effort.The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate.It is a self-assessment scale and is sensitive, reproducible, reliable and validated both in acute pain and chronic pain situations.
Hospitalization lenght (in hours) | 1 week post-surgery
  In case of delayed discharge (the day after the surgery or prolongation of hospitalization), the reasons of prolonged hospital treatment will be collected
Duration of surgical time from the first incision until wound closure (in minutes) | At the moment of wound closure
  Duration of surgical time from the first incision until wound closure will be calculated in minutes
Evolution between inclusion and 24 months post-surgery with regard to quality of life | Inclusion and 1 month post-surgery 12 and 24 months post-surgery
  Quality of life will be assessed using the 36-item Short Form Health Survey (SF-36) score at inclusion and 1 month post-surgery: SF-36 is a standardized and validated questionnaire assessing quality of life. The SF-36 provides two scores: a mental and social quality of life score and a physical quality of life score
The amount of consumed analgesic will be assessed using post-operative data and data reported by the patient on a log book | 7 days post-surgery period
  The amount of consumed analgesic will be measured by calculating the number of patients who have consumed analgesic during the 7 post-operative and antalgic intake (in mg) during the 7 post-operative
Time to return to work or activity post-surgery | Day 1, Day 7 and 1 month post-surgery
  The Time to return to work or activity following surgery will be evaluated in terms of the number of days between hospitalisation and resumption of activity
The rate of early recurrence (at 1 month postoperative) and at long term (12 and 24 months) will be assessed | All study period (24-months)
  Rates of early reccurence during the study (up to one month after surgery). The long-term recurrence rate will also be assessed at 12 and 24 months post-operatively. Recurrence is defined as the reappearance of the hernia on the same side as the one initially operated on, whether the recurrence required surgical intervention.
Number of patients presenting at least one adverse event (AE) | All study period (24-months)
  The safety and tolerability end points will be will be as follows: number of patients presenting at least one adverse event (AE)
Number of patients presenting at least one AE related to the the device implantation | All study period (24-months)
  The safety and tolerability end points will be will be as follows: number of patients presenting at least one AE related to the the device implantation
Number of patients presenting at least one serious adverse event (SAE) | All study period (24-months)
  The safety and tolerability end points will be will be as follows: number of patients presenting at least one serious adverse event (SAE)
Total number of AE related to the device implantation, classified by type and organ | All study period (24-months)
  The safety and tolerability end points will be will be as follows: total number of AE related to the device implantation, classified by type and organ
Satisfaction of the surgeon and unit staff regarding the use of CycloMesh will be evaluated using a satisfaction questionnaire | Day 0
  Surgeon and unit staff will have to answer to a questionnaire concerning the packaging of CycloMesh, the technical characteristics of the implant (flexibility, porosity, etc.), its size, time imbibition of CycloMesh, etc.
Pain intensity after treatment of inguinal hernia by lichtenstein technique under general anesthetic will be assessed 6h post-operative using Visual Analogic Scale (VAS). | 6 hours post-surgery
  The visual analogue scale is a graduated ruler from 0 to 10 cm where 0 indicates that the subject has no pain and 10 cm represents the maximum pain the subject can tolerate. It is a self-assessment scale and is sensitive, reproducible, reliable and validated for both acute and chronic pain situations.
  Pain assessment will be performed 6 hours after implant placement at rest and walking
The rate of patient with chronic pain at 12 and 24 months | 12-months after surgery and 24-months after surgery
  Chronic pain is defined as pain that lasts for at least 6 months after surgery
The rate of implant migration at 12 and 24 months | 12-months after surgery and 24-months after surgery
  Migration is defined as the movement of the entire implant into an organ.
The rate of foreign body sensation at 12 and 24 months postoperative | 12-months after surgery and 24-months after surgery
  Foreign body sensation is assessed by answering yes or no to the question: do you feel a foreign body in the groin

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens Picardie university hospital, Amiens, France